CLINICAL TRIAL: NCT01523483
Title: Vaginal Progesterone for Prevention of Preterm Birth After an Episode of Preterm Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Slovenian Research Agency (Other)
Responsible Party: Principal Investigator, Ziva Novak Antolic, prof. dr. Ziva Novak Antolic, MD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P3-0124
Record Dates: First submitted 2012-01-28; First posted 2012-02-01 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Preterm Birth
Keywords: preterm birth; preterm labor; progesterone; uterine electromyography; cervical length
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progesterone (Experimental): Patients in this arm will receive two micronized progesterone capsules (Utrogestan® 200 mg, i.e. 400 mg of micronized progesterone in sunflower oil) placed into the posterior vaginal fornix once daily for up to 36+6 weeks of gestation.
  Interventions: Drug: Progesterone
- placebo (Placebo Comparator): Patients will receive two placebo capsules placed into the posterior vaginal fornix once daily for up to 36+6 weeks of gestation.
  Interventions: Drug: placebo vaginal capsules

INTERVENTIONS:
Drug: Progesterone — Two micronized progesterone capsules (Utrogestan® 200 mg, i.e. 400 mg of micronized progesterone in sunflower oil) placed into the posterior vaginal fornix once daily for up to 36+6 weeks of gestation.
  Other Names: Brand name: Utrogestan® 200 mg
  Arms: Progesterone
Drug: placebo vaginal capsules — Two placebo capsules placed (soy lecithin and sunflower oil) into the posterior vaginal fornix once daily for up to 36+6 weeks of gestation.
  Arms: placebo

SUMMARY:
The investigators study objective is to investigate the effectiveness of vaginal micronized progesterone in prolonging pregnancy after an episode of preterm labor which responded to tocolytic treatment. Furthermore, the investigators aim is to study the mechanisms of actions of progesterone supplementation by examining its effect on the two components of parturition: cervical ripening and myometrial contractility. The investigators will utilize transvaginal ultrasound to assess the changes in the cervical tissue, and non-invasive trans-abdominal uterine EMG to assess the uterine muscle activity. The investigators will also look at the effect of progesterone on contraction frequency by tocodynamometer (TOCO), though EMG is expected to provide much more information.

ELIGIBILITY:
Inclusion Criteria:

* Patients with singleton pregnancies at gestational ages 25+0 to 33+6 weeks after an episode of preterm labor, with cervical length ≤25mm:
* Patients presenting with signs and symptoms of preterm labor will be admitted and given the standard treatment for preterm labor, i.e. tocolysis for 48 hours, and antenatal steroids.
* Those who will remain undelivered for 48 hours and will be found to have a cervical length of 25mm or less will be offered entrance into the study.
* Preterm labor will be defined as at least 4 contractions in 30 minutes with cervical change assessed by digital cervical examination.

Exclusion Criteria:

* Patients with preterm premature rupture of membranes (PPROM) will be excluded from the study, due to the possibility of ascending infection, as will those with suspected chorioamnionitis.
* We will not include multiple pregnancies.
* Patients with medical conditions that contraindicate tocolysis, such as non-reassuring fetal heart tracings, will also be excluded.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Preterm delivery (before completed 37th week of gestation) | Assessed every 14 days until delivery or 36+6 weeks of gestation

SECONDARY OUTCOMES:
Changes in uterine electromyographic (EMG) activity | Assessed every 14 days until delivery or 36+6 weeks of gestation
  EMG tracing will be analyzed using power density spectrum (PDS) and raw signal amplitude techniques to find mean PDS peak frequency and magnitude. Propagation velocity (PV) of uterine EMG signals will be determined from the time interval between signal arrivals at adjacent electrodes. Amplitude and duration of EMG burst plots will also be analyzed. The study groups will be compared with the PDS, PV and EMG burst plots to determine if progesterone alters the EMG in a way that is less likely to proceed toward labor and delivery.
Cervical length changes | Assessed every 14 days until delivery or 36+6 weeks of gestation
  Cervical length will be measured by transvaginal ultrasound. The study groups will be compared to determine if progesterone alters the cervical shortening process.

CONTACTS AND LOCATIONS:
Overall Officials: Ziva Novak Antolic, PhD, MD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- Univerity Medical Centre Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Background] Lucovnik M, Kuon RJ, Chambliss LR, Maner WL, Shi SQ, Shi L, Balducci J, Garfield RE. Progestin treatment for the prevention of preterm birth. Acta Obstet Gynecol Scand. 2011 Oct;90(10):1057-69. doi: 10.1111/j.1600-0412.2011.01178.x. Epub 2011 Jun 27. PMID 21564026
- [Background] Lucovnik M, Kuon RJ, Chambliss LR, Maner WL, Shi SQ, Shi L, Balducci J, Garfield RE. Use of uterine electromyography to diagnose term and preterm labor. Acta Obstet Gynecol Scand. 2011 Feb;90(2):150-7. doi: 10.1111/j.1600-0412.2010.01031.x. Epub 2010 Dec 7. PMID 21241260
- [Background] Lucovnik M, Maner WL, Chambliss LR, Blumrick R, Balducci J, Novak-Antolic Z, Garfield RE. Noninvasive uterine electromyography for prediction of preterm delivery. Am J Obstet Gynecol. 2011 Mar;204(3):228.e1-10. doi: 10.1016/j.ajog.2010.09.024. Epub 2010 Dec 8. PMID 21145033